CLINICAL TRIAL: NCT02039856
Title: Implementation of VA Womens Health Patient Aligned Care Teams WH-PACTs
Brief Title: Implementation of Women's Health Patient Aligned Care Teams
Acronym: WH-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other); RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CRE 12-026
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Patient-centered Medical Home Implementation
Keywords: Patient-centered medical homes; Primary care; Women's health; Veterans
MeSH Terms: interventions — Quality Improvement; Educational Status

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (cRCT) among 12 VAMCs with unbalanced allocation (2:1) blocked on VA network (Veterans Integrated Service Network or VISN)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBQI-Supported WH-PACT Implementation (Experimental): Evidence-based Quality Improvement (EBQI) is a structured research-clinical partnership approach to facilitating implementation of new care models, including multilevel stakeholder engagement, quality improvement (QI) education/training, technical support, formative feedback, external practice facilitation, and national policy guidance.
  Interventions: Other: Multilevel stakeholder engagement; Other: Quality improvement (QI) education/training; Other: Technical support; Other: Formative feedback; Other: External practice facilitation; Other: National policy guidance
- Routine WH-PACT Implementation (Active Comparator): National policy guidance
  Interventions: Other: National policy guidance

INTERVENTIONS:
Other: Multilevel stakeholder engagement — Structured, in-person stakeholder panel meeting of VA network, VA medical center, and primary care and women's health leaders using modified Delphi panel techniques to come to consensus on a quality improvement (QI) roadmap within each participating VA network, followed by intermittent progress reporting and post-24 months in-person capstone stakeholder panel meetings
  Arms: EBQI-Supported WH-PACT Implementation
Other: Quality improvement (QI) education/training — Initial in-person and ongoing virtual team training in QI principles, methods, and project proposal development and refinement
  Arms: EBQI-Supported WH-PACT Implementation
Other: Technical support — Research team provided technical review of and feedback on local QI project proposals, helped develop and/or recommend process/outcome measures, identified and shared relevant published literature (e.g., measures, interventions), and provided general technical support (e.g., how to analyze local data, how to conduct a local focus group)
  Arms: EBQI-Supported WH-PACT Implementation
Other: Formative feedback — Research team provided aggregated all-site and local data from baseline patient and provider/staff surveys, 12-month patient surveys, and other data and findings to local teams for ongoing and new QI project idea development
  Arms: EBQI-Supported WH-PACT Implementation
Other: External practice facilitation — Within and across site calls with local teams to review progress, identify needs, help solve problems, discuss current and new projects, as well as potential for spread
  Other Names: Facilitation
  Arms: EBQI-Supported WH-PACT Implementation
Other: National policy guidance — VA Handbooks on policy and practice for PACT implementation guidance and on delivery of comprehensive women's health services disseminated to all VA facilities

SUMMARY:
VA has undertaken a major initiative to transform care through implementation of Patient Aligned Care Teams (PACTs). Based on the patient-centered medical home (PCMH) concept, PACT aims to improve access, continuity, coordination and comprehensiveness using team-based care that is patient-driven and patient-centered. However, how VA should adapt PACT to meet the needs of special populations, such as women Veterans, is yet to be worked out. The main goal of this study was to develop and test an evidence-based quality improvement (EBQI) approach to adapting and implementing PACT for women Veterans, incorporating comprehensive women's health care in gender-sensitive care environments, thereby accelerating achievement of PACT tenets for women Veterans and reducing persistent gender disparities in VA quality of care.

DETAILED DESCRIPTION:
Women Veterans' numerical minority in VA healthcare settings has created logistical challenges to delivering gender-sensitive comprehensive services. These challenges only grew as more women Veterans enrolled in VA care. Access and quality lagged behind that of male Veterans, while gender sensitivity, including adequate attention to privacy/safety and awareness of women's military roles and experiences, were often lacking. On-site availability of gender-specific services had also not kept pace, with women Veterans more likely to be outsourced for gender-specific care than they were ten years previously. Further, while the proportion of VA facilities having women's health (WH) clinics had increased, prior research demonstrated that as many as 40% of them were not delivering comprehensive primary care services, instead focusing only on gender-specific exams. Lack of gender-sensitive, comprehensive care for women has also been associated with measurable decrements in women's ratings of VA access, continuity and coordination, as well as measures of technical quality.

The investigators aimed to assess the effectiveness of evidence-based quality improvement (EBQI) methods for developing a WH PACT model using a cluster randomized controlled trial (cRCT) design (Aim #1); examine impacts of receipt of WH-PACT concordant care on women Veterans' outcomes (Aim #2); evaluate processes of EBQI-supported WH-PACT implementation (Aim #3); and develop implementation and evaluation tools for use in EBQI-supported WH-PACT model adaptation, implementation, sustainability and spread to additional VA facilities (Aim #4).

EBQI is a systematic approach to developing a multi-level research-clinical partnership approach to engaging local organizational senior leaders and quality improvement teams in adapting and implementing new care models in the context of prior evidence, local practice context, and provider behavior change methods, with researchers providing technical support and practice facilitation. In a cluster randomized trial, the investigators evaluated WH-PACT model achievement using patient, provider and practice surveys. The investigators examined intermediate changes in provider, staff and team knowledge and attitudes. Using analyses of secondary administrative and performance data, the investigators also explored impacts of receipt of WH-PACT care on quality of chronic disease care and prevention, health status, and utilization. Using mixed methods, the investigators assessed pre-post EBQI practice context; documented WH-PACT implementation; and examined barriers/facilitators to EBQI-supported WH-PACT implementation through a combination of semi-structured interviews and formative progress narratives and administrative data review.

ELIGIBILITY:
Inclusion Criteria:

Facility inclusion criteria:

* VA medical center (VAMC)
* Located in a VISN that has 3 or more VAMCs
* Membership in the Women's Health Practice Based Research Network (PBRN)

Key Stakeholder (interviews) inclusion criteria:

* VISN and VAMC leaders, VAMC primary care/PACT directors, VAMC women's health medical directors, Women Veteran Program Managers (VISN and VAMC), VISN representatives in mental health, health information technology/informatics, quality improvement/system redesign, at least one Nurse Executive (VISN or VAMC)
* Intervention and control VAMCs

Provider (surveys and interviews) inclusion criteria:

* Primary care providers (medical doctor [MD], doctor of osteopathy [DO], nurse practitioner [NP], physician assistant [PA]) who have seen 1+ women Veterans in the past year
* Teamlet primary care provider interviews (MD, DO, NP, PA) at intervention VAMCs
* Surveys of primary care providers (MD, DO, NP, PA) at intervention and control VAMCs
* Surveys of larger primary care/PACT team members (e.g., clinical pharmacists, health coaches)

Staff (surveys and interviews) inclusion criteria:

* Primary care/PACT clinical staff (non-providers) in primary care/PACT teams/teamlets that have seen 1+ women Veterans in the past year
* Teamlet member interviews at Intervention VAMCs

Patient inclusion criteria:

- Women Veterans seen in participating VAMCs with 3+ primary care visits in general primary care and/or women's health clinics in the past year

Exclusion Criteria:

Facility exclusion criteria:

* VA facilities that are not VAMCs (e.g., community-based outpatient clinics or CBOCs)
* VAMCs in VISNs with fewer than 3 VAMCs
* VAMCs that are not members of the WH PBRN

Key Stakeholder (interviews) exclusion criteria:

- Stakeholders outside of the participating VISNs (1, 4, 12, 23) and VAMCs (see study sites)

Provider (surveys and interviews) exclusion criteria:

* VA providers who do not deliver primary care in participating VAMCs
* VA primary care providers who have not seen or do not see women Veteran patients for primary care delivery at a participating VAMC
* Teamlet providers at control VAMCs will not be interviewed

Staff (surveys and interviews) exclusion criteria:

* Primary care clinical staff not participating in PACT (e.g., assigned to primary care rolls but not actually associated with primary care/PACT direct patient care delivery)
* Primary care/PACT clinical staff at control VAMCs will not be interviewed

Patient exclusion criteria:

* Women Veterans who do not use the VA for their health care or for their primary care needs
* Women Veterans with fewer than 3 VA primary care visits in the prior year and therefore not exposed to PACT or WH PACT
* Women Veterans with terminal illness and/or poor prognosis or other health concerns for whom enrollment and survey participation would prove an inappropriate burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only the patient survey component is gender-based (includes women Veterans only). Eligibility for provider/staff surveys or key stakeholder interviews is not gender-based.
Enrollment: 3900 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Yano, PhD MSPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (13):
- United States (13):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Fargo VA Healthcare System, Fargo, ND, Fargo, North Dakota
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Clarksburg Louis A. Johnson VA Medical Center, Clarksburg, WV, Clarksburg, West Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yano EM, Bair MJ, Carrasquillo O, Krein SL, Rubenstein LV. Patient Aligned Care Teams (PACT): VA's journey to implement patient-centered medical homes. J Gen Intern Med. 2014 Jul;29 Suppl 2(Suppl 2):S547-9. doi: 10.1007/s11606-014-2835-8. No abstract available. PMID 24715407
- [Background] Yano EM, Haskell S, Hayes P. Delivery of gender-sensitive comprehensive primary care to women veterans: implications for VA Patient Aligned Care Teams. J Gen Intern Med. 2014 Jul;29 Suppl 2(Suppl 2):S703-7. doi: 10.1007/s11606-013-2699-3. PMID 24715395
- [Result] Chuang E, Brunner J, Mak S, Hamilton AB, Canelo I, Darling J, Rubenstein LV, Yano EM. Challenges with Implementing a Patient-Centered Medical Home Model for Women Veterans. Womens Health Issues. 2017 Mar-Apr;27(2):214-220. doi: 10.1016/j.whi.2016.11.005. Epub 2017 Jan 4. PMID 28063848
- [Result] Hamilton AB, Brunner J, Cain C, Chuang E, Luger TM, Canelo I, Rubenstein L, Yano EM. Engaging multilevel stakeholders in an implementation trial of evidence-based quality improvement in VA women's health primary care. Transl Behav Med. 2017 Sep;7(3):478-485. doi: 10.1007/s13142-017-0501-5. PMID 28585163
- [Result] Goldstein KM, Vogt D, Hamilton A, Frayne SM, Gierisch J, Blakeney J, Sadler A, Bean-Mayberry BM, Carney D, DiLeone B, Fox AB, Klap R, Yee E, Romodan Y, Strehlow H, Yosef J, Yano EM. Practice-based research networks add value to evidence-based quality improvement. Healthc (Amst). 2018 Jun;6(2):128-134. doi: 10.1016/j.hjdsi.2017.06.008. Epub 2017 Jul 13. PMID 28711505
- [Result] Meredith LS, Azhar G, Okunogbe A, Canelo IA, Darling JE, Street AE, Yano EM. Primary Care Providers with More Experience and Stronger Self-Efficacy Beliefs Regarding Women Veterans Screen More Frequently for Interpersonal Violence. Womens Health Issues. 2017 Sep-Oct;27(5):586-591. doi: 10.1016/j.whi.2017.06.003. Epub 2017 Jul 25. PMID 28754476
- [Result] Meredith LS, Wang Y, Okunogbe A, Bergman AA, Canelo IA, Darling JE, Yano EM. Attitudes, Practices, and Experiences with Implementing a Patient-Centered Medical Home for Women Veterans. Womens Health Issues. 2017 Mar-Apr;27(2):221-227. doi: 10.1016/j.whi.2016.11.008. Epub 2017 Jan 10. PMID 28087130
- [Result] Yano EM, Hamilton AB. Accelerating delivery of trauma-sensitive care: Using multilevel stakeholder engagement to improve care for women veterans. Fam Syst Health. 2017 Sep;35(3):373-375. doi: 10.1037/fsh0000288. PMID 28945449
- [Result] Hamilton AB, Yano EM. The importance of symbolic and engaged participation in evidence-based quality improvement in a complex integrated healthcare system: response to "The science of stakeholder engagement in research". Transl Behav Med. 2017 Sep;7(3):492-494. doi: 10.1007/s13142-017-0528-7. PMID 28929322
- [Result] Brunner J, Chuang E, Washington DL, Rose DE, Chanfreau-Coffinier C, Darling JE, Canelo IA, Yano EM. Patient-Rated Access to Needed Care: Patient-Centered Medical Home Principles Intertwined. Womens Health Issues. 2018 Mar-Apr;28(2):165-171. doi: 10.1016/j.whi.2017.12.001. Epub 2018 Jan 12. PMID 29339012
- [Result] Narain K, Bean-Mayberry B, Washington DL, Canelo IA, Darling JE, Yano EM. Access to Care and Health Outcomes Among Women Veterans Using Veterans Administration Health Care: Association With Food Insufficiency. Womens Health Issues. 2018 May-Jun;28(3):267-272. doi: 10.1016/j.whi.2018.01.002. Epub 2018 Feb 21. PMID 29475630
- [Result] Hoggatt KJ, Simpson T, Schweizer CA, Drexler K, Yano EM. Identifying women veterans with unhealthy alcohol use using gender-tailored screening. Am J Addict. 2018 Mar;27(2):97-100. doi: 10.1111/ajad.12689. PMID 29489045
- [Result] Yano EM, Darling JE, Hamilton AB, Canelo I, Chuang E, Meredith LS, Rubenstein LV. Cluster randomized trial of a multilevel evidence-based quality improvement approach to tailoring VA Patient Aligned Care Teams to the needs of women Veterans. Implement Sci. 2016 Jul 19;11(1):101. doi: 10.1186/s13012-016-0461-z. PMID 27435723
- [Result] Brunner J, Cain CL, Yano EM, Hamilton AB. Local Leaders' Perspectives on Women Veterans' Health Care: What Would Ideal Look Like? Womens Health Issues. 2019 Jan-Feb;29(1):64-71. doi: 10.1016/j.whi.2018.10.005. Epub 2018 Nov 16. PMID 30455089
- [Result] Klap R, Darling JE, Hamilton AB, Rose DE, Dyer K, Canelo I, Haskell S, Yano EM. Prevalence of Stranger Harassment of Women Veterans at Veterans Affairs Medical Centers and Impacts on Delayed and Missed Care. Womens Health Issues. 2019 Mar-Apr;29(2):107-115. doi: 10.1016/j.whi.2018.12.002. Epub 2019 Jan 25. PMID 30686577
- [Result] Bergman AA, Hamilton AB, Chrystal JG, Bean-Mayberry BA, Yano EM. Primary Care Providers' Perspectives on Providing Care to Women Veterans with Histories of Sexual Trauma. Womens Health Issues. 2019 Jul-Aug;29(4):325-332. doi: 10.1016/j.whi.2019.03.001. Epub 2019 Apr 23. PMID 31027706
- [Result] Dyer KE, Potter SJ, Hamilton AB, Luger TM, Bergman AA, Yano EM, Klap R. Gender Differences in Veterans' Perceptions of Harassment on Veterans Health Administration Grounds. Womens Health Issues. 2019 Jun 25;29 Suppl 1:S83-S93. doi: 10.1016/j.whi.2019.04.016. PMID 31253247
- [Derived] Yano EM, Than C, Brunner J, Canelo IA, Meredith LS, Rubenstein LV, Hamilton AB. Impact of Evidence-Based Quality Improvement on Tailoring VA's Patient-Centered Medical Home Model to Women Veterans' Needs. J Gen Intern Med. 2024 Jun;39(8):1349-1359. doi: 10.1007/s11606-024-08647-4. Epub 2024 Feb 29. PMID 38424344
- [Derived] Sheahan KL, Goldstein KM, Than CT, Bean-Mayberry B, Chanfreau CC, Gerber MR, Rose DE, Brunner J, Canelo IA, Darling Mshs JE, Haskell S, Hamilton AB, Yano EM. Women Veterans' Healthcare Needs, Utilization, and Preferences in Veterans Affairs Primary Care Settings. J Gen Intern Med. 2022 Sep;37(Suppl 3):791-798. doi: 10.1007/s11606-022-07585-3. Epub 2022 Aug 30. PMID 36042076
- [Derived] Carlson GC, Than CT, Rose D, Brunner J, Chanfreau-Coffinier C, Canelo IA, Klap R, Bean-Mayberry B, Agrawal A, Hamilton AB, Gerber MR, Yano EM. What Drives Women Veterans' Trust in VA Healthcare Providers? Womens Health Issues. 2022 Sep-Oct;32(5):499-508. doi: 10.1016/j.whi.2022.02.004. Epub 2022 Mar 30. PMID 35367107
- [Derived] Danan ER, Brunner J, Bergman A, Spoont M, Chanfreau C, Canelo I, Krebs EE, Yano EM. The Relationship Between Sexual Assault History and Cervical Cancer Screening Completion Among Women Veterans in the Veterans Health Administration. J Womens Health (Larchmt). 2022 Jul;31(7):1040-1047. doi: 10.1089/jwh.2021.0237. Epub 2022 Jan 18. PMID 35049381
- [Derived] Shipherd JC, Darling JE, Klap RS, Rose D, Yano EM. Experiences in the Veterans Health Administration and Impact on Healthcare Utilization: Comparisons Between LGBT and Non-LGBT Women Veterans. LGBT Health. 2018 Jul;5(5):303-311. doi: 10.1089/lgbt.2017.0179. PMID 29979640
- [Derived] Narain K, Jeffers KS, Bean-Mayberry B, Canelo I, Darling JE, Yano EM. The Association of Food Insufficiency with Patient Activation Among Women Veterans Using Veterans Administration Healthcare: a Cross-Sectional Analysis. J Gen Intern Med. 2018 Sep;33(9):1417-1418. doi: 10.1007/s11606-018-4476-9. No abstract available. PMID 29766383
- [Derived] Brunner J, Schweizer CA, Canelo IA, Leung LB, Strauss JL, Yano EM. Timely access to mental health care among women veterans. Psychol Serv. 2019 Aug;16(3):498-503. doi: 10.1037/ser0000226. Epub 2018 Apr 5. PMID 29620391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Random samples of women Veteran clinic users (patient surveys) and census of each VAMC's primary care and women's health providers and staff in PACT and WH-PACT (web surveys) at 12 participating VAMCs recruited through the WH Practice Based Research Network
Units Other Than Participants: VA medical centers
Groups:
- Routine WH-PACT Implementation: PACT implementation is a nationally mandated VA initiative for medical home implementation in VA primary care and women's health clinics, supported by VA Handbooks on PACT and Women's Health policy and practice guidance from national VA primary care and women's health program offices that are disseminated nationally to all VA facilities.
Period: Overall Study
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Started | 2720; 8 VA medical centers | 1180; 4 VA medical centers
Baseline Started - Patients | 2183; 8 VA medical centers | 919; 4 VA medical centers
Baseline Completed - Patients | 953; 8 VA medical centers | 442; 4 VA medical centers
Baseline Started - Providers/Staff | 537; 8 VA medical centers | 261; 4 VA medical centers
Baseline Completed -Providers/Staff | 194; 8 VA medical centers | 94; 4 VA medical centers
Total Baseline Completed | 1147; 8 VA medical centers | 536; 4 VA medical centers
12-month Started-patients | 953; 8 VA medical centers | 442; 4 VA medical centers
12-month Completed- Patients | 580; 8 VA medical centers | 241; 4 VA medical centers
12-month Providers/Staff | 0; 0 VA medical centers | 0; 0 VA medical centers
24-month Started | 1518; 8 VA medical centers | 746; 4 VA medical centers
24-month Started - Patients | 953; 8 VA medical centers | 442; 4 VA medical centers
24-month Completed - Patients | 519; 8 VA medical centers | 222; 4 VA medical centers
24-month Started Providers/Staff | 565; 8 VA medical centers | 304; 4 VA medical centers
24-month Completed Providers/Staff | 174; 8 VA medical centers | 105; 4 VA medical centers
Total 24-month Completed | 693; 8 VA medical centers | 327; 4 VA medical centers
Completed | 693; 8 VA medical centers | 327; 4 VA medical centers
Not Completed | 2027; 0 VA medical centers | 853; 0 VA medical centers
Not completed — Death | 5 | 3
Not completed — Partial survey completion | 61 | 26
Not completed — Lost to Follow-up | 388 | 206
Not completed — Withdrawal by Subject | 1573 | 618

BASELINE CHARACTERISTICS:
Groups:
- Routine WH-PACT Implementation: VA Handbooks on policy and practice for PACT implementation guidance and on delivery of comprehensive women's health services disseminated to all VA facilities
- Total: Total of all reporting groups
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation | Total
Number analyzed (Participants) | 1147 | 536 | 1683
Age, Continuous [Mean (Standard Deviation); unit: years] — Patients only: Age obtained from surveys and VA administrative data during sampling as well as from birth date verified by patients as part of computer-assisted telephone interviews (CATI) Population: There are 4 patients with missing age information, 1 in the EBQI arm and 3 in the control arm.
  years
    Patients: number analyzed (Participants) | 952 | 439 | 1391
    Patients | 53.39 (13.99) | 51.54 (13.76) | 52.80 (13.94)
Age, Customized [Count of Participants; unit: Participants] — Providers/staff only: Age obtained from the surveys Population: There are 27 providers and staff with missing age information; 15 in the EBQI arm and 12 in the control arm.
  Participants
    20-29 years: number analyzed (Participants) | 194 | 94 | 288
    20-29 years | 7 | 3 | 10
    30-39 years: number analyzed (Participants) | 194 | 94 | 288
    30-39 years | 36 | 19 | 55
    40-49 years: number analyzed (Participants) | 194 | 94 | 288
    40-49 years | 48 | 20 | 68
    50-59 years: number analyzed (Participants) | 194 | 94 | 288
    50-59 years | 65 | 30 | 95
    60+ years: number analyzed (Participants) | 194 | 94 | 288
    60+ years | 23 | 10 | 33
    missing: number analyzed (Participants) | 194 | 94 | 288
    missing | 15 | 12 | 27
Sex: Female, Male [Count of Participants; unit: Participants] — Provider/staff specification of sex based on self-report data in web surveys Population: Providers/staff
  Participants
    number analyzed (Participants) | 194 | 94 | 288
    Female | 150 | 72 | 222
    Male | 44 | 22 | 66
Sex: Female, Male [Count of Participants; unit: Participants] — Only female patients were sampled for participation in the computer-assisted telephone interview (CATI) survey using VA administrative data; self-reported sex/gender identity questions were then asked of survey participants. Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    Female | 953 | 442 | 1395
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Providers/staff
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 194 | 94 | 288
    American Indian or Alaska Native | 4 | 0 | 4
    Asian: number analyzed (Participants) | 194 | 94 | 288
    Asian | 7 | 9 | 16
    Black or African American: number analyzed (Participants) | 194 | 94 | 288
    Black or African American | 25 | 11 | 36
    White: number analyzed (Participants) | 194 | 94 | 288
    White | 140 | 55 | 195
    More than one race: number analyzed (Participants) | 194 | 94 | 288
    More than one race | 0 | 1 | 1
    Hispanic or Latino: number analyzed (Participants) | 194 | 94 | 288
    Hispanic or Latino | 4 | 4 | 8
    Unknown or Not Reported: number analyzed (Participants) | 194 | 94 | 288
    Unknown or Not Reported | 18 | 18 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    Asian: number analyzed (Participants) | 953 | 442 | 1395
    Asian | 7 | 3 | 10
    Black or African American: number analyzed (Participants) | 953 | 442 | 1395
    Black or African American | 190 | 129 | 319
    White: number analyzed (Participants) | 953 | 442 | 1395
    White | 630 | 225 | 855
    Hispanic or Latino: number analyzed (Participants) | 953 | 442 | 1395
    Hispanic or Latino | 33 | 37 | 70
    More than one race: number analyzed (Participants) | 953 | 442 | 1395
    More than one race | 83 | 40 | 123
    Unknown or Not Reported: number analyzed (Participants) | 953 | 442 | 1395
    Unknown or Not Reported | 10 | 8 | 18
Post-traumatic stress disorder (PTSD) [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    PTSD positive | 364 | 194 | 558
    PTSD negative | 578 | 244 | 822
    Missing | 11 | 4 | 15
Military Sexual Trauma (MST) [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    MST positive | 575 | 266 | 841
    MST negative | 362 | 167 | 529
    Missing | 16 | 9 | 25
VA care utilization [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    VA-only | 608 | 259 | 867
    VA and non-VA | 345 | 183 | 528
Education [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    Less than college | 180 | 72 | 252
    Some college | 416 | 193 | 609
    College degree | 355 | 176 | 531
    missing | 2 | 1 | 3
Employment [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    Employed | 356 | 193 | 549
    un-employed | 44 | 29 | 73
    Not in labor force | 330 | 125 | 455
    Not in labor force due to disability | 220 | 90 | 310
    missing | 3 | 5 | 8
Stranger harassment from male veterans [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    Never | 737 | 324 | 1061
    Sometimes | 144 | 90 | 234
    Usually | 36 | 14 | 50
    Always | 29 | 13 | 42
    Missing | 7 | 1 | 8
Marital status [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 953 | 442 | 1395
    Single/windowed/divorced/seperated | 573 | 277 | 850
    Married/civil union/ significant other | 371 | 159 | 530
    Missing | 9 | 6 | 15
Are you currently working in WH-PACT? [Count of Participants; unit: Participants] — Population: Providers/staff
  Participants
    number analyzed (Participants) | 194 | 94 | 288
    WH-PACTs | 84 | 27 | 111
    PACTs | 97 | 58 | 155
    not sure | 11 | 5 | 16
    unkown/not reported | 2 | 4 | 6
Proportion of time interacting with patients [Count of Participants; unit: Participants] — Population: Providers/staff
  Participants
    number analyzed (Participants) | 194 | 94 | 288
    1%-24% of my total VA time | 16 | 8 | 24
    25%-49% of my total VA time | 19 | 8 | 27
    50%-75% of my total VA time | 35 | 18 | 53
    >75% of my total VA time | 124 | 60 | 184
Full-time VA employee [Count of Participants; unit: Participants] — Population: Providers/staff
  Participants
    number analyzed (Participants) | 194 | 94 | 288
    Full-time | 178 | 89 | 267
    Part-time | 15 | 5 | 20
    Missing | 1 | 0 | 1
How often do you see or care for women patients in the clinic? [Count of Participants; unit: Participants] — Population: Providers/staff
  Participants
    number analyzed (Participants) | 194 | 94 | 288
    Never | 11 | 10 | 21
    Less than once per month | 57 | 41 | 98
    1-2 times per month | 31 | 7 | 38
    1-2 times per week | 33 | 8 | 41
    several times each week | 20 | 11 | 31
    almost everyday or every day | 40 | 12 | 52
    Missing/not reported | 2 | 5 | 7
Years of service at VA [Mean (Standard Deviation); unit: years] — Population: Providers/staff
  years
    number analyzed (Participants) | 194 | 94 | 288
    (all) | 14.26 (11.77) | 14.75 (10.64) | 14.42 (11.40)

OUTCOME MEASURES:

1. Primary Outcome: WH-PACT Achievement
Description: The Women's Health Patient-Aligned Care Team achievement, based on four patient-reported measures of access to care, patient-provider communication, comprehensiveness of care, and gender-appropriateness of care. The WH-PACT achievement is an aggregate score from -4 to +4, with the higher score meaning better PACT achievement.
Time Frame: Baseline to 24-month
Population: The analysis included the patients who had completed the 24-month survey. One patient in the EBQI arm had missing data for outcome measure and was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 518 | 222
Participants
  Baseline: -4 | 30 | 23
  Baseline: -3 | 49 | 20
  Baseline: -2 | 51 | 26
  Baseline: -1 | 49 | 24
  Baseline: 0 | 59 | 23
  Baseline: +1 | 73 | 31
  Baseline: +2 | 79 | 27
  Baseline: +3 | 75 | 28
  Baseline: +4 | 53 | 20
  24 month: -4 | 34 | 17
  24 month: -3 | 40 | 27
  24 month: -2 | 35 | 15
  24 month: -1 | 41 | 21
  24 month: 0 | 57 | 20
  24 month: +1 | 72 | 24
  24 month: +2 | 93 | 34
  24 month: +3 | 83 | 35
  24 month: +4 | 63 | 29
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in the odds of achieving a higher WH-PACT element; Test type: Superiority — Difference-in-differences using ordered logistic regression, adjusting for age, gender, race/ethnicity, marital status, employment, education, dual use of VA and non-VA for care, diagnosis of PTSD, and the population weights, which were the product of design weights and non-response weights. We verified that proportional odds assumption was met; p = 0.637, difference-in-differences analysis; Odds Ratio (OR) = 0.913, 95% CI 2-sided [0.627 to 1.33], Standard Error of Mean 0.175 — The estimated value is predicted change in the odds of WH-PACT achievement, adjusting for characteristics described in the statistical analysis overview

2. Secondary Outcome: Providers' and Staff Gender Sensitivity
Description: Gender sensitivity score based on 10 survey items related to providers' and staff's sensitivity towards women Veterans during patient care. The score ranged from 1 to 5 with the higher score reflecting greater gender sensitivity toward women Veterans.
Time Frame: Baseline to 24-month
Population: Primary care and women's health providers and staff. The analysis was based on cases with non-missing outcome data. There were 28 missing cases in the EBQI arm and 9 missing in the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EBQI-Supported WH-PACT Implementation: Evidence-based Quality Improvement (EBQI) is a structured research-clinical partnership approach to facilitating implementation of new care models, including multilevel stakeholder engagement, quality improvement (QI) education/training, technical support, formative feedback, external practice facilitation, and national policy guidance.
  Multilevel stakeholder engagement: Structured, in-person stakeholder panel meeting of VA network, VA medical center, and primary care and women's health leaders using modified Delphi panel techniques to come to consensus on a quality improvement (QI) roadmap within each participating VA network, followed by intermittent progress reporting and post-24 months in-person capstone stakeholder panel meetings.
  Quality improvement (QI) education/training: Initial in-person and ongoing virtual team training in QI principles, methods, and project proposal development and refinement
  Technical support: Research team provided technical review of and feedback
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 146 | 96
score on a scale
  Baseline | 4.04 (0.59) | 4.15 (0.57)
  24-month | 4.20 (0.48) | 4.14 (0.62)
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in gender sensitivity score between EBQI and control over time; Test type: Superiority — Difference-in-differences analysis using linear regression, adjusted for gender, race/ethnicity, years worked at VA, worked in women's health clinic vs general primary care clinic, clinician status vs staff status, fulltime employment, percent of women veterans enrolled at the VA facility. We adjusted our analysis using the population weights, which were the product of design weights and non-response weights; p = 0.006, Regression, Linear; Median Difference (Final Values) = 0.33, 95% CI 2-sided [0.10 to 0.57], Standard Error of Mean 0.1195 — The estimated value reported here is the predicted mean change over time, adjusting for characteristics described in the statistical analysis overview

3. Secondary Outcome: Team Functioning
Description: Perceived team functioning of primary care and women's health providers and staff, measured based on responses to 7 survey items. The team functioning score ranged from 1 to 5 , with the higher score indicating better team functioning.
Time Frame: Baseline to 24-month
Population: Primary care and women's health providers and staff. The analysis was based on cases with non-missing outcome data. There are 80 missing cases in the EBQI arm and 74 in the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 94 | 31
score on a scale
  Baseline | 3.70 (0.84) | 4.10 (0.71)
  24 month | 3.84 (0.75) | 3.98 (0.77)
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in team functioning score between EBQI and control over time; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.055, Regression, Linear; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.01 to 0.87], Standard Error of Mean 0.2253 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Providers and Staff Burnout
Description: Burnout was measured using one item: "How often does the following statement apply to you: I feel burned out from my work" with options for 1.Never, 2. A few times a year, 3. Every month, 4. A few times a month, 5. Every week, 6. A few times a week, 7. Every day. We recoded the responses into a binary value: never/less than a few times a month (1-4) and every week-to-everyday (5-7).
Time Frame: 24-month
Population: Primary care and women's health providers and staff. The analysis was based on cases with non-missing burnout data. There were 30 missing cases in the EBQI arm and 10 in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 144 | 95
Participants
  nver/less than a few times a month (1-4) | 112 | 72
  everyweek to everyday (5-7) | 32 | 23
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Test type: Superiority — We adjusted our analysis using the population weights, which were the product of design weights and non-response weights; p = 0.058, Regression, Logistic; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.13 to 1.04], Standard Error of Mean 0.1922 — The estimated value is the predicted mean, adjusting for weights, worked in women's health vs general PC clinic, years worked at the VA, race/ethnicity, gender, full-time employment, and percent of women veterans enrolled at the VA facility

5. Secondary Outcome: Patient VA Primary Care Visits Per Year
Description: Average number of visits to VA primary care per year
Time Frame: Baseline to 24month
Population: Patients only. One patient in the EBQI arm had missing outcome information and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: average visits per year for all patients
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 518 | 222
average visits per year for all patients
  Baseline | 6.96 (5.57) | 6.46 (5.14)
  24month | 6.78 (7.21) | 5.16 (5.90)
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in number of patient primary care visits between EBQI and control over time; Test type: Superiority — Difference-in-differences analysis using linear regression, adjusted for age, gender, race/ethnicity, marital status, employment, education, dual use of VA and non-VA for care, diagnosis of PTSD. We adjusted our analysis using the population weights, which were the product of design weights and non-response weights; p = 0.008, Regression, Linear; Median Difference (Net) = 1.25, 95% CI 2-sided [0.14 to 2.36], Standard Error of Mean 0.56 — The estimated value is predicted change in the number of VA primary care visits, adjusting for characteristics described in the statistical analysis overview

6. Secondary Outcome: Patient VA Women's Health Care Visits Per Year
Description: Average number of patient visits to VA women's health care per year
Time Frame: Baseline to 24month
Population: Patients only. One patient in the EBQI arm had missing outcome information and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Average visits per year for all patients
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 518 | 222
Average visits per year for all patients
  Baseline | 4.05 (4.41) | 4.63 (3.74)
  24month | 4.23 (6.23) | 3.24 (3.69)
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in number of patient visits to women's health care between EBQI and control over time; Test type: Superiority — Difference-in-differences analysis using linear regression, adjusted for adjusted for survey weights, age, gender, race/ethnicity, marital status, employment, education, dual use of VA and non-VA for care, diagnosis of PTSD, and the population weights, which were the product of design weights and non-response weights; p = 0.000, Regression, Linear; Median Difference (Net) = 1.69, 95% CI 2-sided [0.88 to 2.51], Standard Error of Mean 0.413 — The estimated value is predicted change in the number of VA women's health visits, adjusting for characteristics described in the statistical analysis overview

7. Secondary Outcome: Patient VA Hospitalization
Description: Average number of patient hospitalization for any cause in a year
Time Frame: Baseline to 24-month
Population: Patients only. One patient in the EBQI arm had missing outcome information and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Average visits per year for all patients
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 518 | 222
Average visits per year for all patients
  Baseline | 0.26 (0.82) | 0.19 (0.63)
  24-month | 0.17 (0.60) | 0.15 (0.41)
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in number of patient hospitalization for any cause between EBQI and control over time; Test type: Superiority — Difference-in-differences analysis using linear regression, adjusted for adjusted for survey weights, age, gender, race/ethnicity, marital status, employment, education, dual use of VA and non-VA for care, diagnosis of PTSD. We adjusted our analysis using the population weights, which were the product of design weights and non-response weights; p = 0.794, Regression, Linear; Median Difference (Net) = -0.018, 95% CI 2-sided [-0.15 to 0.12], Standard Error of Mean 0.068 — The estimated value is predicted change in the number of VA hospitalization, adjusting for characteristics described in the statistical analysis overview

8. Secondary Outcome: Patient Emergency Room Visits
Description: Average number of patient emergency room visits for any cause in a year
Time Frame: baseline to 24-month
Population: Patients only. One patient in the EBQI arm had missing outcome information and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Average visits per year for all patients
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
Number analyzed (Participants) | 518 | 222
Average visits per year for all patients
  Baseline | 0.90 (1.89) | 0.72 (1.31)
  24-month | 0.78 (1.50) | 0.55 (1.05)
Statistical Analysis 1: Comparison: EBQI-Supported WH-PACT Implementation vs Routine WH-PACT Implementation; Change in number of emergency room visits for any cause between EBQI and control over time; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.888, Regression, Linear; Median Difference (Net) = 0.021, 95% CI 2-sided [-0.265 to 0.306], Standard Error of Mean 0.15 — The estimated value is predicted change in the number of VA emergency room visits, adjusting for characteristics described in the statistical analysis overview

ADVERSE EVENTS:
Time Frame: No adverse events were expected for EBQI-supported WH-PACT implementation (target of action is VA employees). However, we did collect data from women Veteran routine primary care patients. Eligible patients were considered low-risk, so a formal suicidality assessment was not included. However, in an abundance of caution, any survey respondent who endorsed feeling down, depressed or hopeless at baseline, 12-months or 24-months received information about VA's suicide hotline.
Description: Patients were not directly involved in this research other than to participate in a survey.
Groups:
- Routine WH-PACT Implementation: National policy guidance including VA Handbooks on policy and practice for PACT implementation guidance and on delivery of comprehensive women's health services disseminated to all VA facilities.
Arm/Group | EBQI-Supported WH-PACT Implementation | Routine WH-PACT Implementation
All-Cause Mortality (participants affected / at risk) | 5/2720 | 3/1180
Serious Adverse Events (participants affected / at risk) | 0/2720 | 0/1180
Other Adverse Events (participants affected / at risk) | 0/2720 | 0/1180

LIMITATIONS AND CAVEATS:
Control arm VAMCs are active controls given national mandates to implement PACT and WH PACT. Low response rates among providers/staff may have resulted in under- or over-estimation of effects, despite weighting for non-response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT02039856/Prot_SAP_000.pdf